CLINICAL TRIAL: NCT04654910
Title: Does Patient-Reported Outcome Measure Use in Clinic Visits Improve Patient Satisfaction and Experience? A Randomized, Controlled Trial
Brief Title: PROMIS and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Orthopaedic Foot and Ankle Society (Unknown)
Responsible Party: Principal Investigator, Judy Baumhauer, MD, Professor and Associate Chair Orthopaedics, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00005316
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Ankle Pathology; Foot Pathology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): enrolled subjects that do NOT receive explanation of PROMIS measures during visit.
  Interventions: Behavioral: Placebo
- Intervention (Active Comparator): enrolled subjects that DO receive explanation of PROMIS measures during visit.
  Interventions: Behavioral: PROMIS Score Explanation

INTERVENTIONS:
Behavioral: PROMIS Score Explanation — The surgeon completing the clinical visit with the participant will explain what the PROMIS tool is, the purpose of the tool and what the participant's scores mean using a script.
  Arms: Intervention
Behavioral: Placebo — Subjects will complete the PROMIS assessment but will not receive an explanation of the tool.
  Arms: Control

SUMMARY:
The primary aim for this study is to determine if patient satisfaction and experience is improved with the active discussion/inclusion of PROMIS scores during new foot and ankle clinic patient visits.

ELIGIBILITY:
Inclusion

* Patients over the age of 18
* New patient at the foot and ankle clinic

Exclusion

* Patients under the age of 18
* Patients presenting for a Follow up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
mean pain interference domain measured by PROMIS | baseline, before intervention
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Scores are typically between 20-80, but may be 0-100. Any result with higher a higher number is indicating higher pain interference effect.
mean Patient Activation Measure (PAM) | baseline, after intervention
  Our primary outcome measure is the Patient Activation Measure (PAM). The PAM is a 13-item scale with a 5-point Likert response scale for all questions. Raw scores are scaled to a range of 0-100 with 100 being the highest activation in self- management.
percent of participant who respond favorably on the Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG CAHPS) | baseline, after intervention
  We will assess scores on the Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG CAHPS) survey. This is a standardized tool to measure patients' perception of care provided by physicians in an office setting. Specifically, for our analysis will we focus specifically on the individual question to assess communication. We will compare the percentage of participants in the intervention versus control group who respond favorably to this question using a chi-square test of association.
mean depression | baseline, before intervention
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Scores are typically between 20-80, but may be 0-100. Any result with higher a higher number is indicating higher depression effect.
mean physical function | baseline, before intervention
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Scores are typically between 20-80, but may be 0-100. Any result with higher a higher number is indicating higher physical function effect.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
participant data will not be available for other researchers. data is to remain in house at URMC.